CLINICAL TRIAL: NCT01435213
Title: Competition With Striatal [11C]ORM-13070 Binding by Atipamezole and Endogenous Noradrenaline - a PET Study in Healthy Human Subjects
Brief Title: Competition With Striatal [11C]ORM-13070 Binding by Atipamezole and Endogenous Noradrenaline
Acronym: AIMI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Turku (Other)
Collaborators: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Principal Investigator, Juha Rinne, Professor, University of Turku
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: 3099002
Record Dates: First submitted 2011-09-14; First posted 2011-09-16 (Estimated); Last update posted 2013-02-18 (Estimated); Status verified 2013-02

CONDITIONS: Healthy
Keywords: alpha2-adrenoceptor; receptor occupancy; positron emission tomography; [11C]ORM-13070; striatum; brain; noradrenaline; norepinephrine; endogenous; binding; Validation studies
MeSH Terms: interventions — atipamezole; Atomoxetine Hydrochloride; Ketamine; Insulin; insulin, neutral

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (6):
- Atipamezole (Experimental)
  Interventions: Drug: Atipamezole
- Atomoxetine (Experimental)
  Interventions: Drug: Atomoxetine
- Ketamine (Experimental)
  Interventions: Drug: Ketamine
- Insulin-induced hypoglycemia (Experimental)
  Interventions: Drug: Insulin
- Cold pressor test (Experimental)
  Interventions: Other: Cold pressor test
- Placebo (Experimental)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atipamezole — Administration of a single dose of 5-150 micrograms of atipamezole as an intravenous infusion
  Other Names: ANTISEDAN VET
  Arms: Atipamezole
Drug: Atomoxetine — A single dose of 1.2 mg/kg of atomoxetine administered orally
  Other Names: Strattera
  Arms: Atomoxetine
Drug: Ketamine — A single dose of ketamine (approximately 60 mg) administered as an intravenous infusion
  Other Names: Ketalar
  Arms: Ketamine
Other: Cold pressor test — 30-45 min cold pressor test of the foot
  Arms: Cold pressor test
Drug: Insulin — Insulin administered as an intravenous infusion to induce hypoglycemia
  Other Names: Insulin Actrapid
  Arms: Insulin-induced hypoglycemia
Drug: Placebo — A single dose of placebo (capsules) administered orally
  Arms: Placebo

SUMMARY:
The purpose of this study is to validate [11C]ORM-13070 as an alpha2C-adrenoceptor imaging agent for human positron emission tomography (PET) studies of brain alpha2C-adrenoceptor occupancy.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent (IC) obtained.
* Good general health ascertained by detailed medical history, laboratory investigations and physical examination.
* Males between 20 and 40 years of age (inclusive).
* Body mass index (BMI) between 18-28 kg/m2 inclusive (BMI = weight/height2).
* Weight 60-100 kg (inclusive).

Exclusion Criteria:

* Suspected poor compliance with the protocol or inability to communicate well with the study personnel.
* Veins unsuitable for repeated venipuncture.
* CYP2D6 slow metabolizer or ultrarapid metabolizer genotype.
* Evidence of clinically significant cardiovascular, renal, hepatic, haematological, gastrointestinal, pulmonary, metabolic-endocrine, neurological, urogenital or psychiatric disease as judged by the investigator.
* Any condition requiring regular concomitant medication including herbal products or likely to need any concomitant medication during the study.
* Susceptibility to severe allergic reactions.
* Intake of any medication that could affect the outcome of the study, within 2 weeks prior to the tracer administration (2 months for enzyme inducing drugs like rifampicin or carbamazepine), or less than 5 times the half-life of the medication.
* Regular consumption of more than 21 units of alcohol per week (1 unit = 4 cl spirits, about 13 g of alcohol).
* Current use of nicotine-containing products more than 5 cigarettes or equivalent/day.
* Inability to refrain from using nicotine-containing products during the stay at the study centre.
* Inability to refrain from consuming caffeine-containing beverages during the stay at the study centre, e.g. propensity for headache when refraining from caffeine-containing beverages.
* Blood donation or loss of significant amount of blood within 2 months prior to the screening visit.
* Abnormal 12-lead electrocardiogram (ECG) finding of clinical relevance after 10 minutes rest in supine position at the screening visit, for example:
* QTc (calculated using Bazett's formula) > 450 msec,
* PR < 120 msec or > 210 msec,
* QRS < 70 msec or > 120 msec.
* Heart rate (HR) < 40 beats/minute or > 90 beats/minute after 10 minutes rest in supine position at the screening visit.
* At the screening visit, systolic blood pressure (BP) < 90 mmHg or > 140 mmHg after 10 minutes in supine position, diastolic BP < 50 mmHg or > 90 mmHg after 10 minutes in supine position.
* Any abnormal laboratory value, vital sign or physical examination result, which may in the opinion of the investigator interfere with the interpretation of the test results or cause a health risk to the subject if he takes part in the study.
* History of drug abuse or positive result in drug abuse test.
* Positive serology to human immunodeficiency virus antibodies (HIVAb), hepatitis B surface antigen (HBsAg) or hepatitis C virus antibodies (HCVAb).
* Anatomical abnormality in brain MRI which may in the opinion of the investigator interfere with the interpretation of the PET results.
* Any other condition that in the opinion of the investigator would interfere with the evaluation of the results or constitute a health risk to the subject.
* Participation in another clinical drug study within 3 months prior to this study.
* Participation in a prior PET study or other medical or occupational exposure to significant doses of ionizing radiation.
* Any contraindication to MRI of the brain.

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2011-09; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Receptor occupancy | 30 minutes
  PET tracer (interventional drug) uptake in the brain is measured for 30 minutes by PET after various pharmacological and physiological pre-treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Juha Rinne, MD, PhD, Principal Investigator — University of Turku
Locations (2):
- Finland (2):
  - University of Turku, Clinical Research Services Turku CRST, Turku
  - University of Turku, Turku PET Centre, Turku

REFERENCES:
- See also: Clinical Research Services Turku CRST — http://www.crst.fi
- See also: Turku PET Centre — http://www.turkupetcentre.fi/